CLINICAL TRIAL: NCT06889610
Title: A Single-center,Multi-cohort,Prospective Phase II Clinical Study of Multimodal Ablation Combined With Systemic Drug Therapy for Advanced Solid Tumors.
Brief Title: A Phase II Clinical Study of Multimodal Ablation Combined With Systemic Drug Therapy for Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, Chief Physician, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTTP1-DHF-610
Record Dates: First submitted 2025-02-17; First posted 2025-03-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Triple Negative Breast Cancer Metastatic; Melanoma Metastatic; Colorectal Cancer Metastatic
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Experimental): Colorectal Cancer Cohort
  Interventions: Combination Product: MTT(Multimodal Tumor Thermal Therapy System)- Colorectal Cancer
- B (Experimental): Triple-Negative Breast Cancer Cohort
  Interventions: Combination Product: MTT(Multimodal Tumor Thermal Therapy System)- Triple-Negative Breast Cancer
- C (Experimental): Melanoma Cohort
  Interventions: Combination Product: MTT(Multimodal Tumor Thermal Therapy System)- Melanoma

INTERVENTIONS:
Combination Product: MTT(Multimodal Tumor Thermal Therapy System)- Colorectal Cancer — Multimodal ablation combined with cadonilimab and fruquintinib
  Arms: A
Combination Product: MTT(Multimodal Tumor Thermal Therapy System)- Triple-Negative Breast Cancer — Multimodal ablation combined with pucotenlimab and TPC or sacituzumab govitecan, eribulin,gemcitabine,UTD1
  Arms: B
Combination Product: MTT(Multimodal Tumor Thermal Therapy System)- Melanoma — Multimodal ablation combined with pucotenlimab, with other specific agents determined based on the first-line treatment regimen and the melanoma subtype.
  Arms: C

SUMMARY:
This study focuses on the treatment of liver metastases from three common cancers: colorectal cancer, triple-negative breast cancer and melanoma. Currently, there are limitations in the treatment of liver metastases of these cancers. Multimodal thermophysical ablation therapy can reshape the tumor microenvironment, release neoantigens, and act as an in-situ vaccine. On this basis, the combination of multimodal ablation with immunotherapeutic drugs such as pucotenlimab will be explored. The efficacy and safety of this combination therapy in patients with liver metastases of solid tumors will be investigated, with the expectation of breaking through the existing treatment limitations.

ELIGIBILITY:
Inclusion Criteria i. Common eligibility criteria for all cohorts:

1. Age between 18-80 years,gender not limited; 2. The number of liver metastases is≥3.Besides the ablation lesions,there must be at least one measurable lesion(≥1cm),and the diameter of the ablation lesions is<5cm; 3. Expected survival≥3 months; 4. ECOG performance status score of 0-1; 5. Within 14 days before the first dose,laboratory tests indicate adequate organ function:

a) Hematology:WBC≥3.0×10^9/L;ANC≥1.5×10^9/L;PLT≥75×10^9/L;HGB≥90 g/L b) Liver function:Child-Pugh score≤7,AST≤5.0×ULN;ALT≤5.0×ULN;TBIL≤1.5×ULN c) Renal function:Cr≤1.5×ULN or CrCl≥60 mL/min d) Coagulation function:INR≤1.5×ULN(for patients on anticoagulant therapy,≤3×ULN,anticoagulants must be discontinued one week before ablation);APTT≤1.5×ULN ii. Additional eligibility criteria for each cohort:

1. Colorectal Cancer：

   a) Clinically or pathologically confirmed colorectal cancer with liver metastases that are unresectable, or the patient is intolerant to or refuses surgery; b) Patients who have failed standard second-line drug therapy.
2. Triple-negative breast cancer :

   1. Clinically or pathologically confirmed triple-negative breast cancer(triple-negative defined as<1% nuclear staining for ER and PR expression and HER2 negative);
   2. Patients who have failed standard second-line drug therapy(including those who have failed PD-1 monoclonal antibody therapy, with progression within six months of adjuvant or neoadjuvant therapy considered as first-line therapy failure).
3. Melanoma :

   1. Clinically or pathologically confirmed melanoma liver metastasis, with inoperable or intolerable liver lesions or refusal of surgical resection;
   2. Patients who have failed standard first-line drug therapy.

Exclusion Criteria:

i. Common exclusion criteria for all cohorts:

1. Patients with known allergy or suspected allergy to the study drugs or similar drugs;
2. Patients who have participated in another clinical study and received at least one treatment within 4 weeks prior to enrollment;
3. History or concurrent presence of other malignant tumors(except for cured basal cell carcinoma of the skin,superficial bladder cancer,carcinoma in situ of the cervix,and papillary thyroid carcinoma);
4. Patients with immunodeficiency diseases within 7 days prior to the first dose,or currently receiving systemic corticosteroid therapy(≥10mg/day prednisone or equivalent dose of other corticosteroids),or other forms of immunosuppressive therapy;
5. Symptomatic central nervous system(CNS)metastases,or other evidence indicating that the CNS metastases have not been controlled,and deemed unsuitable for enrollment by the investigator;
6. Patients who have previously undergone organ or bone marrow transplantation;
7. Uncontrollable pleural effusion,pericardial effusion,or ascites causing respiratory syndrome(≥CTCAE grade 2 dyspnea);
8. Esophageal(gastric fundus)variceal rupture bleeding within the last month;
9. Other antitumor treatments outside the combined regimen,such as radiotherapy,systemic chemotherapy,etc.;
10. Clinically significant electrolyte abnormalities as judged by the investigator;
11. Insufficiency or failure of major organs;
12. Patients who have received systemic drug therapy,radiotherapy,or local liver treatment,with a time interval of less than 1 month since the last systemic treatment or local liver treatment;
13. Patients who have received immunotherapy and experienced grade 3 or higher immune-related adverse events(irAEs)(except for thyroid function abnormalities,blood sugar abnormalities);
14. Active or uncontrolled severe infections(≥CTCAE grade 2 infections);
15. Any other disease,clinically significant metabolic abnormalities,physical examination abnormalities,or laboratory test abnormalities that,in the investigator's judgment,may have a disease or condition that makes the patient unsuitable for the study drug,or may affect the interpretation of the study results,or may place the patient at high risk;
16. Pregnant or breastfeeding women,or women of childbearing age with a positive baseline pregnancy test;
17. Known human immunodeficiency virus(HIV)infection;known clinically significant liver disease history,including viral hepatitis[known carriers of hepatitis B virus(HBV)must exclude active HBV infection,i.e.,HBV DNA positive(>1×10^4 copies/mL or>2000 IU/mL);known hepatitis C virus(HCV)infection and HCV RNA positive(>1×10^3 copies/mL),or other hepatitis,cirrhosis;
18. Patients with severe heart,lung,liver,or kidney dysfunction,irreversible coagulation disorders,or other uncontrolled diseases(including hypertension or diabetes,active infections,mental illness,or social conditions that may affect patient compliance);
19. Other factors that may affect patient safety or trial compliance as judged by the investigator.

ii. Additional exclusion criteria for each cohort:

1. Colorectal Cancer :

   a) Patients with uncontrolled hypertension, defined as: patients with hypertension that cannot be well-controlled with a single antihypertensive agent (SBP ≥150 mmHg or DBP ≥100 mmHg); or patients who require two or more antihypertensive medications to control blood pressure.

   b）Patients with urine dipstick proteinuria ≥2+ and a 24-hour urinary protein level >1.0 g.

   c）Patients with gastrointestinal diseases such as active gastric or duodenal ulcers, ulcerative colitis, or active bleeding from an unresected tumor; or other conditions judged by the investigator as potentially causing gastrointestinal bleeding or perforation.

   d）Patients with evidence or history of a significant bleeding tendency within 3 months prior to enrollment (e.g., bleeding >30 mL, hematemesis, melena, hematochezia), hemoptysis (>5 mL of fresh blood within 4 weeks), or a thromboembolic event (including stroke and/or transient ischemic attack) within the past 12 months.

   e）Patients with clinically significant cardiovascular disease, including but not limited to, acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months prior to enrollment.

   f）Congestive heart failure of New York Heart Association (NYHA) class > II; ventricular arrhythmias requiring medication; or an ECG showing a QTc interval ≥480 milliseconds.

   g）Patients who are unable to take fruquintinib orally.
2. Triple-negative breast cancer :

   a) Patients who have previously received Pucotenlimab treatment;
3. Melanoma :

   1. Patients who have previously received Pucotenlimab treatment;
   2. Patients currently have uncontrolled hypertension,defined as:patients with hypertension that cannot be well controlled with monotherapy(systolic blood pressure≥150 mmHg,or diastolic blood pressure≥100 mmHg);or patients using two or more antihypertensive drugs to control blood pressure;
   3. Urine routine indicates proteinuria≥2+,and 24-hour urine protein>1.0g;
   4. Significant clinically meaningful cardiovascular diseases,including but not limited to acute myocardial infarction,severe/unstable angina,or coronary artery bypass grafting within 6 months before enrollment;
   5. Congestive heart failure New York Heart Association(NYHA)classification>2;ventricular arrhythmias requiring drug treatment;electrocardiogram(ECG)showing QTc interval≥480 milliseconds.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 2 years.
  It refers to the proportion of patients whose tumors have reduced by a certain amount and maintained for a certain period,including cases of Complete Response(CR)and Partial Response(PR).Objective tumor responses are assessed using the Response Evaluation Criteria in Solid Tumors(RECIST 1.1).Subjects must have measurable tumor lesions at baseline,and the criteria for efficacy assessment are classified according to RECIST 1.1 as Complete Response(CR),Partial Response(PR),Stable Disease(SD),and Progressive Disease(PD).

SECONDARY OUTCOMES:
Disease Control Rate | Up to 2 years.
  It includes the percentage of patients with confirmed cases of Complete Response(CR),Partial Response(PR),and Stable Disease(SD)out of those who are evaluable for efficacy.Subjects must have measurable tumor lesions at baseline,and the criteria for efficacy assessment are classified according to RECIST 1.1 as Complete Response(CR),Partial Response(PR),Stable Disease(SD),and Progressive Disease(PD).
Duration of Response | Up to 2 years.
  The duration of response is defined as the time interval from the start of the response(when CR or PR is first confirmed)to the time of progression or death(whichever occurs first).
Progression-Free Survival | Up to 2 years.
  It refers to the time from the date of enrollment to the date of the first recorded disease progression(PD)or death,whichever occurs first.
Overall Survival | Up to 2 years.
  Overall Survival(OS) refers to the time from the date of enrollment to the date of death due to any cause.
Safety and Tolerability | Up to 2 years.
  Safety refers to the extent to which a drug does not cause unacceptable harm or side effects when applied in the human body.Tolerability refers to the degree to which patients accept the side effects that occur after treatment,reflecting their ability to endure the side effects of the medication.All adverse events will be recorded and assessed for severity based on the NCI-CTC AE 5.0 grading criteria.During the follow-up period,all subjects will be continuously monitored,and the occurrence,duration,severity,and treatment-relatedness of adverse events will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No